CLINICAL TRIAL: NCT04349423
Title: Daily Assessment of Mood and Social Media Behaviors Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-131-ROQA
Record Dates: First submitted 2020-02-19; First posted 2020-04-16 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Anxiety; Stress; Depression; Cortisol
Keywords: Social Media
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to social media usage groups to assess if reduction social media will improve mood and in turn lower depressive and anxiety symptoms. The groups include 0 minutes, 30 minutes, 1 hours of use a day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Social Media Use (Experimental): Participants will be asked to refrain from using all social media
  Interventions: Behavioral: Social Media Usage Manipulation
- Maximum 30 minutes of use (Experimental): Participants will be asked to only use social media at most 30 minutes a day.
  Interventions: Behavioral: Social Media Usage Manipulation
- Maximum 1 hour of use (Experimental): Participants will be asked to only use social media at most 60 minutes a day.
  Interventions: Behavioral: Social Media Usage Manipulation
- Control (Experimental): Control Group
  Interventions: Behavioral: Social Media Usage Manipulation

INTERVENTIONS:
Behavioral: Social Media Usage Manipulation — Behavioral Intervention of social media usage.

SUMMARY:
The purpose of this research study is to learn more about social media usage and its relation to emotions, biology, and mental health. Participants will complete daily assessments (5 times a day) over the course of 11 days in which they will report on their social media use, behaviors, and mood. During the first 4 days participants will be asked to continue using social media as typical. In the second half (7 days) participants will be randomized to social media usage groups (0 minutes, 30 minutes, 1 hour, 2 hour, 3 hours). There will be mental health and well-being measures provided at the beginning and end of the study. Lastly, to better understand how social media usage effects underlying mechanisms of stress, participants will be asked to provide saliva samples for 3 nights (pre, mid, and post) to assess for basal cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Having a smartphone

Exclusion Criteria:

* Below age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in "Positive and Negative Affect Schedule" (PANAS) | Pre and post. Daily 5 times a day for 11 days
  Examines mood fluctuations. Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Changes in "Depression Anxiety and Stress Scale" (DASS) | Pre and Post. Daily for 11 days
  Examines Depressive, Anxiety, and Stress symptoms. Minimum 0 maximum 63. Higher scores indicate more depression, anxiety and or stress.
Changes in "Behavioral Activation for Depression Scale" | Pre-Post- Daily for 11 days
  Examines behavioral goal achievement. Minimum 0 and maximum 54. Larger scores means an ability to be more active.
Changes in "Social Media Use" | Daily for 11 days
  Survey and Phone based Applications will assess for daily use of social media time and behaviors.
Changes in "A clinically useful depression outcome scale" (CUDOS) | Pre-Post- Daily for 11 days
  Tracks Depression Symptoms. Minimum 0 maximum 74. Larger scores means more depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Methodist University, Dallas, Texas, United States